CLINICAL TRIAL: NCT00299377
Title: Randomized Comparison of Abciximab i.v. Versus i.c. in Primary PCI Patients With STEMI and Effects on Infarct Size and Microvascular Obstruction
Brief Title: Abciximab i.v. Versus i.c. in Primary PCI Patients With STEMI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Leipzig (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-Thiele
Record Dates: First submitted 2006-03-02; First posted 2006-03-06 (Estimated); Last update posted 2008-07-03 (Estimated); Status verified 2008-06

CONDITIONS: Myocardial Infarction
Keywords: STEMI; infarct size; primary PCI; no-reflow; ST-elevation myocardial infarction
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction

INTERVENTIONS:
Drug: Abciximab i.v.
Drug: Abciximab i.c.

SUMMARY:
Randomized comparison of abciximab i.v. versus i.c. in patients with STEMI undergoing primary PCI. The hypothesis is, that higher concentration of abciximab i.c. leads to improved epicardial flow, perfusion, reduction of no-reflow, reduction in infarct size and subsequently better outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical symptoms:

   * Angina < 12 h persistent Angina > 30 min.
2. ECG-Criteria:

   * ST-elevation > 1mm in ≥ 2 extremity leads
   * ST-elevation > 2mm in ≥ 2 contiguous anterior leads
3. Informed consent

Exclusion Criteria:

1. No consent
2. Pregnancy
3. Allergy against abciximab, ASA or heparin
4. Active peptic ulcus ventriculi or duodeni
5. Active non-superficial bleeding
6. Major surgical intervention, intracerebral interventions, puncture central artery < 4 weeks
7. Active internal bleeding
8. Cerebrovascular complications < 2 years
9. Known coagulation disorders, thrombocytopenia
10. Arteriovenous malformations or aneurysms
11. Severe Liver or renal dysfunction
12. Severe untreated hypertension
13. Active vasculitis
14. Previous thrombolysis < 12 h

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2006-01; Primary Completion 2007-11; Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Infarct size and microvascular obstruction assessed by MRI

SECONDARY OUTCOMES:
ST-segment resolution, TIMI-Flow, TIMI blush grade, ejection fraction, left ventricular volumes, clinical outcome (MACE)

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, Principal Investigator — Heart Center Leipzig - University Hospital
Locations (1):
- University of Leipzig - Heart Center, Leipzig, Germany

REFERENCES:
- [Derived] de Waha S, Desch S, Eitel I, Fuernau G, Zachrau J, Leuschner A, Gutberlet M, Schuler G, Thiele H. Impact of early vs. late microvascular obstruction assessed by magnetic resonance imaging on long-term outcome after ST-elevation myocardial infarction: a comparison with traditional prognostic markers. Eur Heart J. 2010 Nov;31(21):2660-8. doi: 10.1093/eurheartj/ehq247. Epub 2010 Jul 30. PMID 20675660
- [Derived] Thiele H, Schindler K, Friedenberger J, Eitel I, Furnau G, Grebe E, Erbs S, Linke A, Mobius-Winkler S, Kivelitz D, Schuler G. Intracoronary compared with intravenous bolus abciximab application in patients with ST-elevation myocardial infarction undergoing primary percutaneous coronary intervention: the randomized Leipzig immediate percutaneous coronary intervention abciximab IV versus IC in ST-elevation myocardial infarction trial. Circulation. 2008 Jul 1;118(1):49-57. doi: 10.1161/CIRCULATIONAHA.107.747642. Epub 2008 Jun 16. PMID 18559698